CLINICAL TRIAL: NCT02287766
Title: Prognostic Indicators for Metabolic Syndrome as Provided by the EPIC ClearView
Brief Title: Metabolic Syndrome Feasibility Study
Acronym: EPIC-009
Status: Completed | Type: Observational
Sponsor: Epic Research & Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EPIC-009
Record Dates: First submitted 2014-11-05; First posted 2014-11-11 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control: Men and women ages 21-85 lacking any medical diagnosis (as defined in the protocol) of one or more of the following cancer, coronary artery disease or heart attack, renal failure or dialysis, hepatitis, Multiple Sclerosis, or any autoimmune disorder.
- Metabolic Syndrome Diagnosis Group: Men and women ages 21-85 with at least of at least three of the following (as defined in the protocol) : Elevated waist circumference, elevated triglycerides, reduced HDL cholesterol, elevated blood pressure, elevated fasting glucose.

SUMMARY:
The objective of this study is to determine whether the finger tip images captured by the EPIC ClearView device, when analyzed via the ClearView software, produce a Response Scale that characterizes trends consistent with Metabolic Syndrome identified by medical doctors.

ELIGIBILITY:
Metabolic Group

Inclusion Criteria:

1. Sex: Male or Female
2. Age range: 21 to 85
3. Qualifying Metabolic Syndrome diagnosis(using the National Cholesterol Education Program Adult Treatment Panel (ATP) III definition)(Grundy, 2004)

   Subjects will be identified as having Metabolic Syndrome if they meet at least three of the following five criteria:
   * Elevated waist circumference: ≥ 102 cm (≥40 inches) in men, ≥ 88 cm (≥35 inches) in women
   * Elevated triglycerides: ≥ 150 mg/dL (1.7 mmol/L) or on drug treatment for elevated triglycerides (examples include, but are not limited to, fibrates and nicotinic acid)
   * Reduced HDL cholesterol: < 40 mg/dL (1.03 mmol/L) in men or < 50 mg/dL (1.3 mmol/L) in women or on drug treatment for reduced HDL-C
   * Elevated blood pressure: ≥ 130 mm Hg systolic blood pressure or ≥85 mm Hg diastolic blood pressure or on antihypertensive drug treatment in a patient with a history of hypertension
   * Elevated fasting glucose: ≥ 100 mg/dL or on drug treatment for elevated glucose
4. The patient or legal representative is able to understand and provide signed consent for the procedure.

Exclusion Criteria:

1. Patients < 21years in age or > 85 years in age.
2. Inability or unwillingness to provide informed consent.
3. Patients with pacemakers or another electrical device implanted somewhere in their body.
4. Pregnant women.
5. Missing all or part of fingers or cuts/burns on pads of fingers
6. Hand tremors or involuntary oscillations of the hands that prevents clear imaging

Control Group:

Inclusion Criteria:

1. Sex: Male or Female
2. Age range: 21 to 85
3. Freedom from qualifying medical diagnoses (control group)

Any one of the following will exclude the subject from participation in the study

1. Documented current diagnosis/treatment of cancer (including Sickle Cell Disease)
2. Documented current diagnosis/treatment of coronary artery disease or heart attack
3. Documented as currently in Renal Failure (chronic or acute) or on renal dialysis
4. Documented current diagnosis/treatment for Hepatitis

5 .The patient or legal representative is able to understand and provide signed consent for the procedure.

Exclusion Criteria:

1. Patients < 21 years in age or > 85 years in age.
2. bility or unwillingness to provide informed consent.
3. Patients with pacemakers or another electrical device implanted somewhere in their body.
4. Pregnant women.
5. Missing all or part of fingers or cuts/burns on pads of fingers
6. Hand tremors or involuntary oscillations of the hands that prevents clear imaging

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men and women ages 21-85 who present to the investigators clinical office and meet all of the inclusion criteria while having none of the exclusion criteria will be approached for consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Agreement of ClearView Scan versus Active Diagnosis | At time of ClearView Scan (Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit
  The EPIC ClearView software produces a Response Scale report that summarizes the electrophysiological measurements associated with organ systems. The autonomic numbers indicate how the person's stress response is affecting different body systems and the physical numbers reflect physiological function.These measurements will then be compared to metabolic diagnosis.

SECONDARY OUTCOMES:
Sensitivity and Specificity of ClearView Scan versus Active Diagnosis | Single study visit only, with no follow-up. The study endpoint will be reported for day 0, the day of the study visit

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Rizzo, PhD, Principal Investigator — EPIC Research and Diagnostics
Locations (2):
- United States (2):
  - EPIC Research and Diagnostics, Scottsdale, Arizona
  - Integrated Health Institute, LLC, Scottsdale, Arizona